CLINICAL TRIAL: NCT00334048
Title: Treatment of Sexual Dysfunction Secondary to Antidepressant Pharmacotherapy: A Double-blind Comparison of Requip (Ropinirole) vs. Placebo in Patients Taking SSRI Antidepressants
Brief Title: Treating Sexual Dysfunction From Selective Serotonin Reuptake Inhibitor (SSRI) Medication: a Study Comparing Requip CR to Placebo
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St. Luke's-Roosevelt Hospital Center (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: David J. Hellerstein, MD, NY State Psychiatric Institute
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 06-036; NYSPI IRB# 5185
Record Dates: First submitted 2006-06-02; First posted 2006-06-06 (Estimated); Last update posted 2015-02-19 (Estimated); Status verified 2015-02

CONDITIONS: Sexual Dysfunction
Keywords: Medication-induced sexual dysfunction; SSRI-induced sexual dysfunction; Anorgasmia; Delayed ejaculation; Sexual dysfunction; Antidepressant-induced sexual dysfunction; Requip; Ropinirole; Dopamine agonist; Serotonin reuptake inhibitor; Sexual dysfunction, physiological, medication-induced
MeSH Terms: conditions — Sexual Dysfunction, Physiological; Ejaculatory Dysfunction | interventions — ropinirole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Ropinirole (Requip) — 1 mg extended release formulation given once per day to a maximum of 4 per day
  Other Names: requip, ropinirole, requip XL

SUMMARY:
Antidepressant medicines sometimes cause sexual side effects. The purpose of this study is to determine whether the sexual dysfunction sometimes caused by selective serotonin reuptake inhibitor (SSRI) antidepressant medications can be reversed by treatment with Requip (ropinirole), a medicine which is used to treat Parkinson's Disease and restless leg syndrome.

DETAILED DESCRIPTION:
A significant proportion of patients taking pharmacotherapy for treatment of depression experience sexual dysfunction at distressing levels, with reported rates varying considerably. When sexual dysfunction is assessed prospectively using structured questionnaires, high levels of dysfunction have been found. SSRIs including paroxetine, sertraline, and other medications, have been shown to have a similar frequency of sexual side effects and in a recent prospectively designed study 50% of men taking sertraline reported that they were only "slightly" (18%) or "not at all" (32%) satisfied with their sexual functioning. It is reported that sexual side effects of antidepressant treatment frequently result in noncompliance with and/or premature discontinuation of treatment. A recent study showed that the dopamine agonist Requip (Ropinirole) reduced the amount of SSRI-associated sexual dysfunction. The proposed study will utilize a placebo control group in a crossover design to determine the effect on sexual dysfunction of adding Requip (Requip CR formulation) to the patient's SSRI treatment.

30 patients experiencing sexual dysfunction attributable to SSRI treatment for depression will be entered into this study. All patients will receive 6 weeks of treatment with Ropinirole and 6 weeks with placebo in a crossover fashion. Assessments of sexual functioning and depression will be made at each visit.

ELIGIBILITY:
Inclusion Criteria:

1. male or female outpatients 18-65 years old
2. currently taking fluoxetine, sertraline, paroxetine, citalopram, or escitalopram at a stable dosage within the ranges specified for 1 month or longer required dosage range: (Prozac (fluoxetine) 20-80 mg/day; Celexa (citalopram) 20-60 mg/day; Lexapro (escitalopram) 10-30 mg/day; Zoloft (sertraline) 50-200 mg/day; Paxil (paroxetine) 20-60 mg/day; Paxil CR (paroxetine CR) 25-75 mg/day
3. Currently responding to the SSRI antidepressant treatment, as indicated by

   * a score of 15 or less on the HDRS 24 item at screening and baseline, and (b) CGI-Severity score of 2 or less at baseline
4. Meets DSM-IV criteria for Substance-Induced Sexual Dysfunction, with impairment of desire, arousal, or orgasm
5. Are currently involved in an intimate relationship which includes sexual contact
6. agree to use double-barrier contraception during sexual intercourse during the course of the study (women only)
7. Agree to the study team contacting the physician who prescribe their SSRI medication to inform them of their participation in the current study

Exclusion Criteria:

1. Patients with a DSM-IV diagnosis of Delirium, Dementia, and Amnestic, and other Cognitive Disorders,
2. Patients with a principal diagnosis meeting DSM-IV criteria for: Bipolar Disorder or cyclothymia, Schizophrenia, Delusional (Paranoid) Disorders and Psychotic Disorders Not Otherwise Specified, or Anorexia Nervosa or Bulimia,
3. Patients who, within the past 6 months, met DSM-IV criteria for abuse of or dependence on any drug, including alcohol,
4. Patients who would pose a serious risk for suicide during the course of the study, as evidenced by one of the following:

   * report of having a specific plan for killing themselves,
   * a score of 3 or higher on the Hamilton Depression Rating Scale item 3 as rated by the study doctor at the first visit, (indicative of active suicidal thoughts or behaviors), or
   * a suicide attempt within the past 6 months,
5. Patients with a history of medical conditions or procedures which may cause sexual dysfunction, including: peripheral vascular disease, radical prostatectomy, trans-urethral resection of the prostate [TURP], or spinal cord injury.
6. History of sexual dysfunction predating onset of depression and/or initiation of antidepressant therapy,
7. Patients receiving any other treatment for sexual dysfunction, including sex therapy
8. Pregnant or nursing women.
9. Patients with unstable or life-threatening medical conditions, such as uncontrolled hypertension, diabetes, or hypothyroidism, acute infections, pneumonia, severe renal or hepatic impairment.
10. Patients with any the following: retinal disease, sleep apnea, or narcolepsy.
11. Patients taking dopamine agonist medication.
12. Patients taking medications that are

    * associated with orthostatic hypotension, such as tricyclic antidepressants, MAO Inhibitors, and alpha1 antagonists
    * CYP1A2 inhibitors, such as fluoroquinolones, fluvoxamine, cimetidine
    * SSRI medication used cyclically for PMDD
13. Patients who do not expect to have regular sexual contact with another person over the next 13 weeks.
14. Patients with a DSM-IV diagnosis of Pathological Gambling

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2006-06; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
International Index of Erectile Function (IIEF) | 6 weeks
Sexual Function and Satisfaction Questionnaire (SFSQ) | 6 weeks

SECONDARY OUTCOMES:
Hamilton Depression Rating Scale, 17 items (HDRS-17) | 6 weeks
Global Assessment of Functioning Scale (GAFS) | 6 weeks
Clinical Global Impressions (CGI) | 6 weeks
CGI-Sexual functioning (CGI-Sx) | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David J. Hellerstein, MD, Principal Investigator — St. Luke's Roosevelt Hospital Center and NY State Psychiatric Institute
Locations (1):
- Mood Disorders Research Program, New York, New York, United States

REFERENCES:
- [Background] Worthington JJ 3rd, Simon NM, Korbly NB, Perlis RH, Pollack MH; Anxiety Disorders Research Program. Ropinirole for antidepressant-induced sexual dysfunction. Int Clin Psychopharmacol. 2002 Nov;17(6):307-10. doi: 10.1097/00004850-200211000-00006. PMID 12409684
- [Background] Balon R. Sexual function and dysfunction during treatment with psychotropic medications. J Clin Psychiatry. 2005 Nov;66(11):1488-9. doi: 10.4088/jcp.v66n1120. No abstract available. PMID 16420088
- See also: Mood Disorders Research Program website — http://www.depressionny.com
- See also: Columbia Psychiatry website — http://www.columbiapsychiatry.org/research/clinics/mdrp.html